CLINICAL TRIAL: NCT00531167
Title: Prospective Randomized Study for the Comparison of Adding Adefovir Dipivoxil and Switching to Entecavir in Patients With Lamivudine-resistant Chronic Hepatitis B
Brief Title: Adding Adefovir Dipivoxil Versus Switching to Entecavir in Patients With Lamivudine-resistant Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Hyung Joon Yim, associate professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRT 111098
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Hepatitis B
Keywords: lamivudine resistant mutations; rescue therapy
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; adefovir dipivoxil; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): combination therapy
  Interventions: Drug: combination of lamivudine+adefovir vs entecavir
- B (Active Comparator): entecavir
  Interventions: Drug: combination of lamivudine+adefovir vs entecavir

INTERVENTIONS:
Drug: combination of lamivudine+adefovir vs entecavir — Lamivudine 100 mg/day, Adefovir 10 mg/day, Entecavir 0.5 mg/day
  Other Names: Zeffix, Hepsera, Baraclude

SUMMARY:
Antiviral resistance mutations limit the efficacy of therapy for chronic hepatitis B. At year 2, resistance to adefovir may occur as high as 25% in patients with history of lamivudine resistance. Resistance to entecavir is reported to be 10% in lamivudine refractory patients during the same period. However, combination of lamivudine and adefovir decreased the adefovir resistance rate as low as 0% in the recent studies. By overcoming the antiviral resistance, the efficacy of therapy will be maximized. This study is intended to compare the efficacy of two strategies, combination of lamivudine and adefovir vs. entecavir monotherapy in patients with lamivudine resistance.

DETAILED DESCRIPTION:
Recently, published data showed combination of lamivudine and adefovir lead to PCR negativity (<1000 copies/mL) up to 80% in the treatment of lamivudine-resistant chronic hepatitis B at year 2 [Rapti et al. Hepatology 2007 Feb;45(2):307-13.]. Other studies also showed 76% and 69% PCR negativity in mostly HBeAg negative subjects [Lampertico et al. Hepatology 2006 Oct;44(4) Suppl 1:556A-557A, Lampertico et al. Hepatology 2006 Oct;44(4) Suppl 1:693A-694A].

In the study for the treatment of lamivudine-resistant chronic hepatitis B patients which included HBeAg positive subjects more predominantly, entecavir monotherapy showed 34% of PCR negativity (<300 copies/mL) at year 2 [Tenney DJ, et al. Antimicrob Agents Chemother. 2007 Mar;51(3):902-11].

Although it is assumed that combination of lamivudine and adefovir would be more effective than entecavir monotherapy for lamivudine resistant patients, we cannot verify the assumption, because there is no data directly comparing these two strategies until now.

The aim of this study is to determine the most effective therapy for the patients with lamivudine resistant chronic hepatitis B. We will compare the PCR negativity (<60 IU/ml) of HBV DNA at year 2 in patients receiving 'the combination of lamivudine and adefovir' and 'entecavir monotherapy'.

Since we are planning to include lamivudine-resistant chronic hepatitis B patients regardless of HBeAg status, we assumed the PCR negativity (<300 copies/mL or <60 IU/mL) in adefovir-lamivudine combination and entecavir monotherapy group as 55% and 34%, respectively, considering HBeAg status and lower detection limit of PCR.

The result of this study will be able to clearly demonstrate the superiority of combination therapy with lamivudine and adefovir to entecavir monotherapy, which provide us the guide to rescue therapy for patients with lamivudine resistant HBV.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic hepatitis B patients (positive HBsAg > 6 months)
2. Age > 16 year old
3. Serum alanine aminotransferase (ALT) >1.5 x ULN
4. History of treatment with lamivudine more than 6 months
5. Proven lamivudine resistant mutation
6. HBV DNA level> 20000 IU/mL
7. Compensated liver disease (Child-Pugh-Turcotte score over 7; prothrombin time prolonged more than 3 sec above ULN or INR over 1.5; serum albumin >3 g/dL; total bilirubin <2.5 mg/dL; No history of variceal bleeding, ascites, or hepatic encephalopathy)
8. Patients willing to give informed consent

Exclusion Criteria:

1. Out of inclusion criteria
2. Any one of following

   * Serum phosphorus level under 2.4 mg/dL
   * Serum creatinine level over 1.5 mg/dL or creatinine clearance <50 mL/min
   * Absolute neutrophil count lower than 1000 cell/mL
   * Hb level under 10 g/dL (male), under 9 g/dL (female)
   * Serum AFP >100 ng/mL
3. History of treatment with interferon-a, thymosin-alfa 1, or nucleos(t)ide analogue other than lamivudine in 6 months of screening
4. Recipient of organ transplantation
5. Positive antibody test to HIV, HCV or HDV
6. Pregnant or breast feeding women
7. Patients with hepatocellular carcinoma or uncontrolled malignant disease
8. Habitual alcohol drinker (>140 g/week for men, >70 g/week for women)

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
PCR negativity (<60 IU/ml) of HBV DNA | At the end of year 2 (since starting rescue therapy for lamivudine resistance)

SECONDARY OUTCOMES:
1. PCR negativity (<60 IU/ml) of HBV DNA at year 1 (interim analysis) 2. Degrees of HBV DNA reduction 3. ALT normalization 4. HBeAg seroconversion 5. Development of resistant mutation 6. Virologic breakthrough 7. Biochemical breakthrough | At the end of year 2 except interim analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Joon Yim, M.D., Principal Investigator — Korea University; Eileen Yoon, Study Director — Korea University; Yeon Seok Seo, M.D, Study Director — Korea University; Soon Ho Um, M.D, Study Director — Korea University; Chang Wook Kim, M.D, Study Director — The Catholic University of Korea; Chang Don Lee, Study Director — The Catholic University of Korea; Sang Hoon Park, M.D, Study Director — Hallym University; Myung Seok Lee, M.D, Study Director — Hallym University; Choong Kee Park, M.D, Study Director — Hallym University; Hee Bok Chae, M.D, Study Director — Chungbuk National University; Moon young Kim, M.D, Study Director — Yonsei University; Soon Koo Baik, M.D, Study Director — Yonsei University; Ju Hyun Kim, M.D, Study Director — Gachon University Gil Medical Center; Yun Soo Kim, M.D, Study Director — Gachon University Gil Medical Center; Jung Il Lee, M.D, Study Director — Inha University; Jin Woo Lee, M.D, Study Director — Inha University; Sun Pyo Hong, PhD, Study Director — Genematrix Inc.
Locations (2):
- South Korea (2):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Korea University Anam Hospital, Seoul

REFERENCES:
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B. Hepatology. 2007 Feb;45(2):507-39. doi: 10.1002/hep.21513. No abstract available. PMID 17256718
- [Background] Rapti I, Dimou E, Mitsoula P, Hadziyannis SJ. Adding-on versus switching-to adefovir therapy in lamivudine-resistant HBeAg-negative chronic hepatitis B. Hepatology. 2007 Feb;45(2):307-13. doi: 10.1002/hep.21534. PMID 17256746
- [Background] Tenney DJ, Rose RE, Baldick CJ, Levine SM, Pokornowski KA, Walsh AW, Fang J, Yu CF, Zhang S, Mazzucco CE, Eggers B, Hsu M, Plym MJ, Poundstone P, Yang J, Colonno RJ. Two-year assessment of entecavir resistance in Lamivudine-refractory hepatitis B virus patients reveals different clinical outcomes depending on the resistance substitutions present. Antimicrob Agents Chemother. 2007 Mar;51(3):902-11. doi: 10.1128/AAC.00833-06. Epub 2006 Dec 18. PMID 17178796
- [Background] Peters MG, Hann Hw Hw, Martin P, Heathcote EJ, Buggisch P, Rubin R, Bourliere M, Kowdley K, Trepo C, Gray Df Df, Sullivan M, Kleber K, Ebrahimi R, Xiong S, Brosgart CL. Adefovir dipivoxil alone or in combination with lamivudine in patients with lamivudine-resistant chronic hepatitis B. Gastroenterology. 2004 Jan;126(1):91-101. doi: 10.1053/j.gastro.2003.10.051. PMID 14699491